CLINICAL TRIAL: NCT05260918
Title: Understanding Physiology of Float-REST and the Consequential Effects on Subjective and Objective Recovery in Individuals With Chronic Lower Back Pain
Brief Title: Examining the Effects of Float-REST for Recovery in Individuals With Chronic Lower Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West Virginia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2010130921
Record Dates: First submitted 2022-01-13; First posted 2022-03-02 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-05

CONDITIONS: Pain, Chronic
Keywords: Sensory Deprivation Tank; fMRI
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flotation-REST (Active Comparator): Float-REST therapy uses sensory deprivation tanks that consist of a very large warm water enclosure with a high concentration of Epsom salt to create a completely buoyant environment. This, along with a combination of temperature that is kept equal to skin temperature (94 degrees), allows the participant to eliminate the gravitational effects on the body, and along with lack of sound and low to no light (depending on comfort) allows the brain and body to completely relax for augmented physical and mental recovery. The room will contain an intercom that allows participants to communicate with study personnel in the event the participant needs assistance. Participants will undergo 60 minute sessions twice a week for 3 weeks.
  Interventions: Other: Float-REST
- Nappod (Placebo Comparator): Participants in this arm will be asked to lie comfortably in a special recliner called a Metro Nappod for the duration of a 60 minute session twice a week for 3 weeks. The chair is located in a quiet and dimly lit room to minimize interruptions. The pod is equipped with a privacy visor, built-in speaker, and a timer with an alarm.
  Interventions: Other: Nappod

INTERVENTIONS:
Other: Float-REST — Participants will utilize sensory deprivation tanks.
  Arms: Flotation-REST
Other: Nappod — Participants will utilize nappod.
  Arms: Nappod

SUMMARY:
Researchers at the West Virginia University Rockefeller Neuroscience Institute are looking for volunteers to participate in a research study to evaluate what effects Float-REST (Restricted environmental Stimulation Technique) has on the stress response caused by chronic lower back pain.

DETAILED DESCRIPTION:
Chronic lower back pain has a profound impact on a patient's life and body. These patients face a litany of internal and external stressors. These stressors cause a detrimental sustained activation of the endogenous stress response, which is mediated by the autonomic nervous system. Our central hypothesis is that this high stress load exacerbates the symptoms of chronic pain by causing changes in how the brain processes pain signals from the periphery. If researchers can better understand how stress plays a role in the mitigation of pain, then there may be improvements in patient's quality of life. Restricted Environmental Stimulation Therapy (REST) flotation has been identified as a possible alternative treatment to pharmacological intervention for several conditions like generalized anxiety disorder by helping to reduce stress. However, there have yet to be any investigation into what affects that REST flotation has in chronic lower back pain.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to give informed consent
* Right-hand dominant
* Naïve to mindfulness interventions (i.e. guided meditation, guided yoga, previous REST flotation)
* Have chronic lower back pain (at least 12 weeks since onset)
* Ability to enter/exit REST Flotation Tank unassisted
* Stable prescription medication (No changes in dose, start/stop within 30 days of the beginning of the study)

Exclusion Criteria:

* MRI incompatibility: The participant cannot have any non-MRI compatible metallic (magnetic) material in, on, or attached to their body.
* Current fear of small spaces or water
* Current balance problems or motion sickness
* Body width greater than 60cm
* Current contagious skin condition

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-02-24 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Changes in Functional Magnetic Resonance Imaging (fMRI) | Participants will undergo an fMRI session at the beginning (Week 1) to establish a baseline and a follow up end of the study (Week 8).
  fMRI analysis looks at alterations in brain activity from baseline at rest and in response to pain cues

SECONDARY OUTCOMES:
Change in Nocturnal Heart Rate as measured by OURA Ring | Daily from baseline through study completion at 8 weeks
  Heart rate (beats per minute) will be quantified throughout the night via the OURA ring.
Change in daily self-report measures for task load | Daily from baseline through study completion at 8 weeks
  End of Day Questionnaire (EoD)-Developed at the Rockefeller Neuroscience Institute (RNI) as a modification of the NASA Task Load Index. There are 5 Likert scales to assess workload (0=very low and 100=very high), as well as 4 follow up questions. This questionnaire addresses subjective measures of workload and stressors that were encountered throughout the day.
Change in per session self-report measures | Before and after each float session (Weeks 2-7)
  State-Trait Anxiety Index (STAI) - Commonly used measure of state and trait anxiety, and done with 20 very brief questions. Values range from 20 to 80, with higher scores representing more severe anxiety. Participants will complete the STAI questionnaire before and after each session, twice a week.
Change in testing battery self-report measures in personality | Beginning and end of the investigation (Week 1 & Week 8)
  Big Five Inventory (BFI)-44 item inventory designed to measure the Big Five Factors of personality on a 5-point Likert Scale. Higher scores indicate a higher tendency for that personality trait (1=disagree strongly to 5=agree strongly).
Change in testing battery self-report measures in emotional regulation | Beginning and end of the investigation (Week 1 & Week 8)
  Emotion Regulation Questionnaire (ERQ)-10-item scale designed to measure tendency to regulate emotions. Each item is answered on a 7-point Likert Scale (1=strongly disagree to 7=strongly agree). Higher scores indicate a higher emotion regulation strategy.
Change in testing battery self-report measures in mindfulness | Beginning and end of the investigation (Week 1 & Week 8)
  Five Facet Mindfulness Questionnaire (FFMQ)-39 item inventory assesses the five facets of mindfulness on a 5-point Likert Scale (1=never or very rarely true and 5=very often or always true). Each facet is tallied and the sum total responses are divided by 39 (number of items). Higher scores indicate higher levels of mindfulness.
Change in testing battery self-report measures in sleep quality | Beginning and end of the investigation (Week 1 & Week 8)
  Pittsburgh Sleep Quality Index (PSQI)- 19 item inventory with 7 subjective components that assess sleep quality over time. Each component is scored from 0 to 3 (0=very good and 3=very bad). The sum of the components is the global score and ranges 0-21 (0=no difficulty and 21=severe difficulties). The higher the global score, the poorer the sleep quality.
Cold Pressor Stressor | The participant will undergo the cold pressor test at the beginning (Week 1) and end of the study (Week 8) with the option for an additional session after a few sessions at the investigators discretion.
  The cold pressor is a water bath with its temperature maintained at 3C. The participant is asked to submerge a hand in the water bath. The water is cold enough to be a painful stimuli but not so cold as to cause tissue damage. The participant rates their pain level on a standard Wong-Baker pain scale prior and immediately after voluntary withdraw from the cold pressor. The Wong Baker pain scale asks the participant to rate their pain on a scale of 0-10 with 0= no pain and 10= the most pain. Duration of time spent in the water is also recorded.
Serum Analysis for changes in Interleukin 1B concentration | Beginning (Week 1), middle (Week 5), and end of the investigation (Week 8)
  Blood samples will be collected through out the study and analyzed for a key stress indicators Interleukin 1B.
Serum Analysis for changes in Interleukin 6 concentration | Beginning (Week 1), middle (Week 5), and end of the investigation (Week 8)
  Blood samples will be collected through out the study and analyzed for a key stress indicators Interleukin 6.
Serum Analysis for changes in Cortisol concentration | Beginning (Week 1), middle (Week 5), and end of the investigation (Week 8)
  Blood samples will be collected through out the study and analyzed for a key stress indicator Cortisol.
Changes in Serum Analysis for changes in Dehydroepiandrosterone concentration | Beginning (Week 1), middle (Week 5), and end of the investigation (Week 8)
  Blood samples will be collected through out the study and analyzed for a key stress indicator Dehydroepiandrosterone.

CONTACTS AND LOCATIONS:
Overall Officials: Victor S Finomore, PhD, Principal Investigator — West Virginia University
Locations (1):
- Rockefeller Neuroscience Institute at West Virginia University, Morgantown, West Virginia, United States